CLINICAL TRIAL: NCT07061301
Title: Transition to Hospital Discharge in Insulinized Patients With Type 2 Diabetes Mellitus and Incorporation Into a Comprehensive Diabetes Management System
Brief Title: Transition to Hospital Discharge in Insulinized Patients With Type 2 Diabetes Mellitus
Acronym: TRANHOSPIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Principal Investigator, Juan Francisco Merino Torres, Chief of Endocrinology, Professor of Medicine, and Principal Investigator, Instituto de Investigacion Sanitaria La Fe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0338-1
Record Dates: First submitted 2025-05-22; First posted 2025-07-11 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Continuous Glucose Monitoring; CGM; Transition to Discharge; Smart Insulin Pen Cap
Keywords: Type 2 Diabetes Mellitus; cgm; Continuous glucose monitoring; Transition to discharge; smart insulin pen cap; discharge; Insulinized patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This is a pilot, randomized, open-label, parallel-group, single-center clinical trial. Adults with type 2 diabetes who start insulin therapy during hospitalization are randomized prior to discharge into two arms. The intervention group uses a real-time continuous glucose monitor (CGM) and Insulclock® smart cap, while the control group uses both blinded CGM and blinded Insulclock® smart cap and adjusts insulin based on capillary glucose tests. Both groups are followed for 12 weeks with scheduled visits at weeks 1, 2, 4, 8, and 12. The study evaluates adherence to insulin therapy and glycemic control during the hospital discharge transition period. Data are collected digitally in an electronic CRD. Glycemic control is assessed using time in range (TIR), time below range (TBR), time above range (TAR), coefficient of variation, mean glucose, and HbA1c.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Use of blind continuous glucose sensor and smart insulin pen cap. (Active Comparator): From discharge, use of a blind continuous glucose sensor and a smart insulin pen cap. Insulin therapy decision-making based on capillary blood glucose.
  Interventions: Device: Usual Care group
- Use of continuous glucose sensor and smart insulin pen cap and is able to see the parameters. (Experimental): From discharge, a continuous glucose sensor and smart insulin pen cap are used, and the subject is able to see its parameters. Insulin therapy decision-making is based on the continuous glucose sensor and smart cap parameters.
  Interventions: Device: Technological group

INTERVENTIONS:
Device: Usual Care group — Participants will use the same CGM and Insulclock® devices, but in blinded mode (no data available to the patient). Insulin therapy will be adjusted using capillary blood glucose measurements (4 times daily). Device data will be collected retrospectively but not used for treatment decisions.
  Arms: Use of blind continuous glucose sensor and smart insulin pen cap.
Device: Technological group — Participants will use a real-time continuous glucose monitoring device (e.g., FreeStyle Libre 2) and the Insulclock® smart insulin pen cap. Both devices provide real-time feedback and data on insulin administration and glucose levels. Patients will adjust their insulin therapy based on these data.
  Arms: Use of continuous glucose sensor and smart insulin pen cap and is able to see the parameters.

SUMMARY:
This clinical study explores whether adding technological tools during hospital discharge can help people with type 2 diabetes who are starting insulin therapy achieve better treatment adherence and blood glucose control once they return home. The discharge transition period includes both the final days of hospitalization and the first weeks to months after returning home.

When people with type 2 diabetes are hospitalized, they sometimes need to begin insulin therapy. After discharge, managing insulin properly is essential to avoid high or low blood sugar levels. However, many patients forget or delay insulin doses, which can lead to poor control of their diabetes.

This study will compare two groups of patients. All participants will be adults with type 2 diabetes, between 18 and 70 years old, who are newly starting insulin during their hospital stay.

Group 1 ("technological group") will use a continuous glucose monitor (CGM) and a smart insulin pen cap called Insulclock. These tools show real-time blood glucose data and record when and how much insulin is injected. Patients and doctors can use this information to better adjust treatment. Insulclock also includes alarms to remind patients of their doses.

Group 2 ("control group") will use the same devices, but they will not see the data in real time. Instead, they will manage their insulin based on standard finger-prick blood sugar checks four times a day, as typically done in standard care.

Both groups will be followed for 12 weeks after hospital discharge. Medical check-ins will occur in weeks 1, 2, 4, 8, and 12. Blood tests and treatment adjustments will be performed as needed.

The main goals are:

To measure if the use of technology helps patients stick to their insulin schedule (fewer missed or mistimed injections).

To see if it leads to better blood glucose control (e.g., more time within the recommended range, fewer episodes of low or high glucose).

To evaluate patient satisfaction with this technology and check if the number of unplanned hospital readmissions decreases.

The study will take place at Hospital Universitari i Politècnic La Fe in Valencia, Spain. Around 80 patients will participate.

This study is important because real-world data about the use of CGM and smart insulin devices during the hospital-to-home transition are limited. It may help improve diabetes care for people starting insulin after hospitalization.

DETAILED DESCRIPTION:
The transition from hospital to home is a clinically vulnerable phase for patients with type 2 diabetes mellitus (T2DM), particularly for those who are newly initiated on insulin therapy during hospitalization. This period is characterized by increased therapeutic complexity, limited patient confidence with insulin use, and heightened risk of poor glycemic outcomes. Suboptimal adherence to insulin regimens-including missed or delayed doses-is common and has been associated with adverse clinical events, reduced quality of life, and higher healthcare utilization, including unplanned readmissions.

While continuous glucose monitoring (CGM) systems and smart insulin pen caps have individually shown promise in improving glycemic control and treatment adherence, there is a lack of robust data regarding their effectiveness when introduced in the peri-discharge period. Importantly, the transition from inpatient to outpatient care has been highlighted as a critical moment to implement structured, technology-supported interventions aimed at improving self-management and continuity of care.

This study investigates whether the combination of CGM and Insulclock® technology, initiated during hospitalization and continued after discharge, improves glycemic control and adherence in insulin-treated T2DM patients. Unlike prior studies, this trial evaluates these devices not only as monitoring tools but also as real-time decision-making supports during a period of high clinical risk.

In addition to assessing standard glycemic metrics - including time in range (TIR), time below and above range (TBR, TAR), coefficient of variation, and HbA1c - the study will measure patient-reported treatment satisfaction and unplanned hospital readmissions within 30 days. The outcomes of this research may inform future protocols for diabetes discharge planning and support the integration of connected technologies into standard care pathways for insulin initiation in hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 70 years.
* Hospitalized patients with a diagnosis of type 2 diabetes mellitus (T2DM), either newly diagnosed during admission or previously known but not previously treated with insulin.
* Initiation of insulin therapy (basal, basal-plus, or basal-bolus regimen) during hospitalization, with planned continuation post-discharge.
* Independent in basic activities of daily living.
* Adequate cognitive and functional capacity to manage the required devices: insulin pen, glucometer, continuous glucose monitoring (CGM) sensor, and Insulclock® cap.

Exclusion Criteria:

* Dependence in basic activities of daily living.
* Any medical condition or functional limitation precluding the use of the CGM or the Insulclock® system.
* Pregnancy or intention to become pregnant.
* Diagnosis of type 1 diabetes mellitus.
* Patients undergoing dialysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Therapeutic adherence | From baseline (hospital discharge) to 12 weeks post-discharge
  Assessment of therapeutic adherence based on the number of injustified insulin administration omissions per week. Measured by Number of missed basal and bolus insulin doses within any 14-day period during follow-up.
  Method of Assessment: Data will be collected through the digital insulin pen smart cap system (Insulclock®), which automatically records each insulin administration and detects missed doses.
Time in Range | From baseline (hospital discharge) to 12 weeks post-discharge
  Percentage of time that interstitial glucose values remain within the target range of 70 to 180 mg/dL, as measured by continuous glucose monitoring (CGM). This metric reflects the effectiveness of glycemic control in patients with type 2 diabetes. TIR is widely recognized as a clinically meaningful outcome in diabetes technology studies.
  Unit of Measurement: Percentage (%) of time in target range Method of Assessment: data will be collected from continuous glucose monitoring systems (e.g., Dexcom G6 or equivalent), which record interstitial glucose every 5 minutes. TIR will be calculated over the monitoring period using standard CGM metrics, following international consensus guidelines.
  Justification: TIR has been endorsed as a key metric in diabetes management by the International Consensus on Time in Range. It correlates with reduced risk of microvascular complications and complements traditional measures such as HbA1c.

SECONDARY OUTCOMES:
Time Below Range | From baseline (hospital discharge) to 12 weeks post-discharge
  Percentage of time that interstitial glucose values are below the target range (<70 mg/dL), as measured by continuous glucose monitoring (CGM). TBR will be subdivided into:
  Time in level 1 hypoglycemia: 54-69 mg/dL
  Time in level 2 hypoglycemia: <54 mg/dL
  These thresholds align with the International Consensus on Time in Range.
  Unit of Measurement: Percentage (%) of time below range
  Method of Assessment:
  Data will be extracted from CGM devices (DEXCOM ONE +). The percentage of time spent below each threshold will be calculated using validated software platforms following consensus CGM data analysis protocols.
Time Above Range | From baseline (hospital discharge) to 12 weeks post-discharge
  Percentage of time that interstitial glucose values are above the target range (>180 mg/dL), as measured by CGM. TAR will be subdivided into:
  Time in level 1 hyperglycemia: 181-250 mg/dL
  Time in level 2 hyperglycemia: >250 mg/dL
  Unit of Measurement:
  Percentage (%) of time above range
  Method of Assessment:
  Data will be extracted from CGM device (DEXCOM ONE +). The percentage of time spent above each threshold will be calculated using validated software platforms following consensus CGM data analysis protocols.
Coefficient of Variation | From baseline (hospital discharge) to 12 weeks post-discharge
  The coefficient of variation (CV) of interstitial glucose values over the monitoring period. CV represents glycemic variability and is calculated as the ratio of the standard deviation to the mean glucose level, expressed as a percentage.
  Unit of Measurement:
  Percentage (%)
  Method of Assessment:
  Calculated automatically from CGM data using standard formula: CV = (SD / Mean) × 100. The value will be derived from at least 10 days of valid CGM data, in line with consensus guidelines.
Mean Glucose Level | From baseline (hospital discharge) to 12 weeks post-discharge
  Average interstitial glucose level (mg/dL) measured over the CGM monitoring period. This reflects overall glycemic exposure during the follow-up.
  Unit of Measurement:
  Milligrams per deciliter (mg/dL)
  Method of Assessment:
  Mean glucose will be calculated from CGM recordings collected over the study period, requiring at least 70% device wear-time for valid analysis.
Glycated Hemoglobin (HbA1c) | At 12 weeks post-discharge
  Measurement of glycated hemoglobin (HbA1c), which reflects the average blood glucose concentration over the previous 2-3 months. HbA1c is a standard laboratory marker used to assess long-term glycemic control in patients with diabetes.
  Unit of Measurement:
  Percentage (%)
  Method of Assessment:
  HbA1c will be obtained through standard blood analysis performed during hospitalization and at the 12-week follow-up visit.
Health-related quality of life assessed using the EQ-5D-5L (EuroQol) | At 12 weeks post-discharge
  Assessment of patient health-related quality of life. It will be assessed using the EQ-5D-5L (EuroQol). Outcomes will include the EQ-5D-5L index value derived from the 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and the EQ visual analogue scale (EQ V
  Unit of measurement EQ-5D-5L index value (unitless score) EQ visual analogue scale (EQ VAS), points (0-100)
  Method of assessment Self-administered EQ-5D-5L questionnaire, including 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) with 5 levels each, and the EQ VAS. Higher scores indicate better perceived health status.
Re-hospitalization Rate | Within 30 days post-discharge
  Evaluation of the rate of unplanned hospital readmissions within 30 days following hospital discharge. A sub-analysis will be conducted to classify readmissions based on whether the primary cause was diabetes-related (e.g., hypoglycemia, hyperglycemia, diabetic complications) or non-diabetes-related.
  Unit of Measurement:
  Percentage (%) of participants experiencing hospital readmission.
  Method of Assessment:
  Hospital readmission data will be obtained through review of electronic health records and patient interviews. Only unplanned hospitalizations will be included; planned admissions (e.g., scheduled procedures) will be excluded.
Number of off-schedule insulin administrations | From hospital discharge to 12 weeks post-discharge
  Evaluation of the number of insulin doses administered outside the recommended time window. This includes basal insulin doses administered more than 60 minutes later than scheduled and bolus insulin doses administered more than 15 minutes after the start of the meal. This outcome reflects deviations from the prescribed insulin timing and may indicate suboptimal treatment adherence or workflow issues.
  Unit of Measurement:
  Number of delayed insulin doses per participant
  Method of Assessment:
  Data will be obtained from a connected insulin pen device (Insulclock®), which automatically logs the date and time of each insulin administration. Meal times and prescription schedules will be recorded to determine whether each dose was administered on time or delayed.
Number of participants with abnormal laboratory tests results | During index hospitalization (baseline) and 12 weeks post-discharge
  Several analytical parameters will be assessed in the participants and reported in the Outcome Measure results data table. Blood and urine samples will be collected and analyzed in certified clinical laboratories using standard methods. The following parameters will be measured:
  Blood parameters (units):
  Fasting glucose: mg/dL
  Uric acid: mg/dL
  GGT: U/L
  Total cholesterol: mg/dL
  HDL cholesterol: mg/dL
  LDL cholesterol: mg/dL
  Triglycerides: mg/dL
  ALT (GPT): U/L
  AST (GOT): U/L
  Sodium: mEq/L
  Potassium: mEq/L
  Chloride: mEq/L
  Estimated glomerular filtration rate (eGFR): mL/min/1.73m²
  Creatinine: mg/dL
  Albumin: g/dL
  Glycated hemoglobin (HbA1c): %
  C-peptide: ng/mL
  FIB-4 index: unitless
  Urine parameters:
  Albumin-to-creatinine ratio (ACR): mg/g creatinine
  Urine culture: positive / negative (qualitative)
Use of corticosteroids during hospitalization | During hospitalization (baseline)
  Description:
  Assessment of whether the patient received systemic corticosteroids at any point during the index hospitalization.
  Unit of Measurement:
  Yes / No
  Method of Assessment:
  Information will be obtained from the electronic medical record.
Use of corticosteroids at discharge | At hospital discharge to 12 weeks post-discharge
  Assessment of whether the patient was prescribed systemic corticosteroids at the time of hospital discharge.
  Unit of Measurement:
  Yes / No
  Method of Assessment:
  Information will be obtained from the hospital discharge summary in the electronic medical record.
Insulin dose intensity at discharge | Baseline
  Assessment of total daily insulin dose prescribed at discharge, categorized as ≥0.5 or <0.5 units/kg/day.
  Unit of Measurement:
  Dichotomous: ≥0.5 units/kg/day vs. <0.5 units/kg/day
  Method of Assessment:
  Total daily insulin dose and patient body weight will be extracted from the medical record to calculate the units per kilogram per day.
Insulin dose intensity 12 weeks post-discharge | 12 weeks post-discharge
  Assessment of total daily insulin dose prescribed at 12 weeks post-discharge, categorized as ≥0.5 or <0.5 units/kg/day.
  Unit of Measurement:
  Dichotomous: ≥0.5 units/kg/day vs. <0.5 units/kg/day
  Method of Assessment:
  Total daily insulin dose and patient body weight will be extracted from the medical record to calculate the units per kilogram per day.
Length of hospital stay | During hospitalization
  Duration of the index hospitalization, expressed in total number of days from admission to discharge.
  Unit of Measurement:
  Number of days
  Method of Assessment:
  Calculated from hospital admission and discharge dates recorded in the electronic medical record.
Use of oral antidiabetic drugs at discharge | at hospital discharge and at 12 weeks post-discharge
  Assessment of whether the patient was prescribed any oral antidiabetic medication at the time of hospital discharge. In addition to the yes/no categorization, the specific type(s) of oral antidiabetic agents prescribed (e.g., metformin, DPP-4 inhibitors, SGLT2 inhibitors, sulfonylureas, etc.) will also be recorded.
  Unit of Measurement:
  Yes / No; plus descriptive list of prescribed agents
  Method of Assessment:
  Data will be obtained from the discharge medication list recorded in the electronic medical record. The presence or absence of oral antidiabetic therapy will be noted, along with the names of the active substances prescribed.
Body Weight | Baseline (hospitalization) and at 12 weeks post-discharge
  Measurement of body weight taken with a calibrated scale during hospitalization (baseline) and at 12 weeks post-discharge to assess changes in body composition.
  Unit of Measurement:
  Kilograms (kg)
  Method of Assessment:
  Weight will be measured using a calibrated digital scale at both time points.
Height | Baseline (hospitalization)
  Measurement of participant height to calculate body mass index and assess baseline anthropometrics.
  Unit of Measurement:
  Meters (m)
  Method of Assessment:
  Height will be measured using a stadiometer at enrollment.
Body Mass Index (BMI) | Baseline (hospitalization) and at 12 weeks post-discharge
  Calculation of body mass index (BMI) using weight and height measured at baseline.
  Unit of Measurement:
  Kilograms per square meter (kg/m²)
  Method of Assessment:
  BMI will be calculated as weight (kg) divided by height squared (m²)
Global cardiovascular risk category | Baseline (hospitalization)
  Categorization of participants into global cardiovascular risk groups according to clinical criteria defined in the 2019 ESC/EAS Guidelines for the Management of Dyslipidaemias. Risk levels are determined without the use of SCORE or SCORE2 equations, based on comorbidities, lipid levels, blood pressure, diabetes duration, kidney function, and the presence of established cardiovascular disease or target organ damage.
  Unit of Measurement:
  Categorical: Low / Moderate / High / Very high
  Method of Assessment:
  Participants will be classified into one of four risk categories:
  Very high risk: Established cardiovascular disease, chronic kidney disease stage IV (eGFR <30 mL/min), diabetes with target organ damage or ≥3 major cardiovascular risk factors, or long-standing type 1 diabetes (>20 years)
  High risk: Diabetes duration ≥10 years or with additional risk factors, familial hypercholesterolemia without organ damage, chronic kidney disease stage III
Medication adherence assessed by the 4-item Morisky-Green test (MMAS-4) | At 12 weeks post-discharge
  Brief description Medication adherence assessed using the 4-item Morisky-Green test (MMAS-4).
  Unit of measurement Morisky-Green adherence classification (complier vs non-complier).
  Method of assessment Self-reported 4-item Morisky-Green questionnaire (yes/no responses). Participants are classified as adherent (complier) when all responses indicate adherence; otherwise, they are classified as non-adherent (non-complier).

CONTACTS AND LOCATIONS:
Overall Officials: JUAN FRANCISCO MERINO TORRES, Medicine, Principal Investigator — IIS La Fe; DARIO LARA GALVEZ, Medicine, Study Chair — IIS La Fe; MATILDE RUBIO ALMANZA, Medicine, Study Chair — IIS La Fe
Locations (1):
- Hospital La Fe, Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tian T, Aaron RE, Seley JJ, Longo R, Nayberg I, Umpierrez GE, Levy CJ, Klonoff DC. Use of Continuous Glucose Monitors Upon Hospital Discharge of People With Diabetes: Promise, Barriers, and Opportunity. J Diabetes Sci Technol. 2024 Jan;18(1):207-214. doi: 10.1177/19322968231200847. Epub 2023 Oct 2. PMID 37784246
- [Background] Peyrot M, Barnett AH, Meneghini LF, Schumm-Draeger PM. Insulin adherence behaviours and barriers in the multinational Global Attitudes of Patients and Physicians in Insulin Therapy study. Diabet Med. 2012 May;29(5):682-9. doi: 10.1111/j.1464-5491.2012.03605.x. PMID 22313123
- [Background] Robinson S, Newson RS, Liao B, Kennedy-Martin T, Battelino T. Missed and Mistimed Insulin Doses in People with Diabetes: A Systematic Literature Review. Diabetes Technol Ther. 2021 Dec;23(12):844-856. doi: 10.1089/dia.2021.0164. Epub 2021 Oct 26. PMID 34270324
- [Background] Tejera-Perez C, Chico A, Azriel-Mira S, Lardies-Sanchez B, Gomez-Peralta F; Area de Diabetes-SEEN. Connected Insulin Pens and Caps: An Expert's Recommendation from the Area of Diabetes of the Spanish Endocrinology and Nutrition Society (SEEN). Diabetes Ther. 2023 Jul;14(7):1077-1091. doi: 10.1007/s13300-023-01417-1. Epub 2023 May 15. PMID 37188930
- [Background] Galindo RJ, Ramos C, Cardona S, Vellanki P, Davis GM, Oladejo O, Albury B, Dhruv N, Peng L, Umpierrez GE. Efficacy of a Smart Insulin Pen Cap for the Management of Patients with Uncontrolled Type 2 Diabetes: A Randomized Cross-Over Trial. J Diabetes Sci Technol. 2023 Jan;17(1):201-207. doi: 10.1177/19322968211033837. Epub 2021 Jul 22. PMID 34293955
- [Background] Vinagre I, Mata-Cases M, Hermosilla E, Morros R, Fina F, Rosell M, Castell C, Franch-Nadal J, Bolibar B, Mauricio D. Control of glycemia and cardiovascular risk factors in patients with type 2 diabetes in primary care in Catalonia (Spain). Diabetes Care. 2012 Apr;35(4):774-9. doi: 10.2337/dc11-1679. Epub 2012 Feb 16. PMID 22344609